CLINICAL TRIAL: NCT04643132
Title: S-ketamine Prevents Tibial Fracture-associated Postoperative Pain and Cognitive Dysfunction After Orthopedic Surgery in Patients: a Randomized Double-blind Controlled Trial
Brief Title: S-ketamine Prevents Postoperative Pain and Cognitive Dysfunction After Tibial Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang011
Record Dates: First submitted 2020-11-17; First posted 2020-11-24 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain; Postoperative Cognitive Dysfunction
Keywords: S-ketamine; tibial fracture; orthopedic surgery; pain intensity
MeSH Terms: conditions — Pain, Postoperative; Postoperative Cognitive Complications; Tibial Fractures; Pain | interventions — Saline Solution; Sodium Chloride; Esketamine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal saline in patients (Placebo Comparator): After the induction of anesthesia, normal saline is intravenously injected in a volume of 2ml, and then a continuous infusion of 20 ml/h normal saline until starting skin suture.
  Interventions: Drug: Normal saline
- S-ketamine at low dose in patients (Active Comparator): After the induction of anesthesia, S-ketamine is intravenously injected at 0.2mg/kg, and then a continuous infusion of 0.2mg/kg/h S-ketamine until starting skin suture.
  Interventions: Drug: S-ketamine (low-dose)
- S-ketamine at high dose in patients (Active Comparator): After the induction of anesthesia, S-ketamine is intravenously injected at 0.4mg/kg, and then a continuous infusion of 0.4mg/kg/h S-ketamine until starting skin suture.
  Interventions: Drug: S-ketamine (high-dose)

INTERVENTIONS:
Drug: Normal saline — After the induction of anesthesia, normal saline is intravenously injected in a volume of 2ml, and then a continuous infusion of 20ml/h normal saline until starting skin suture.
  Other Names: 0. 9% Sodium Chloride Injection
  Arms: Normal saline in patients
Drug: S-ketamine (low-dose) — After the induction of anesthesia, S-ketamine is intravenously injected at 0.2mg/kg, and then a continuous infusion of 0.2mg/kg/h S-ketamine until starting skin suture.
  Other Names: Esketamine Hydrochloride Injection
  Arms: S-ketamine at low dose in patients
Drug: S-ketamine (high-dose) — After the induction of anesthesia, S-ketamine is intravenously injected at 0.4mg/kg, and then a continuous infusion of 0.4mg/kg/h S-ketamine until starting skin suture.
  Other Names: Esketamine Hydrochloride Injection
  Arms: S-ketamine at high dose in patients

SUMMARY:
Purpose:

To explore effects of S-ketamine on postoperative pain and cognitive dysfunction after tibial fracture and orthopedic surgery.

To evaluate and examine the incidence of adverse effects with the purpose of selecting the optimum dose.

DETAILED DESCRIPTION:
With the increase in human life span, orthopedic injuries and subsequent repair surgery have become a major health problem which impairs the life quality of patients and burdens healthcare systems worldwide. Poor post-surgical pain control is a leading factor that hinders the physical rehabilitation and musculoskeletal functional recovery, and causes acute cognitive impairment and chronic pain syndrome. Also, existing treatments of opioids and non-steroidal anti-inflammatory drugs have potential drawbacks, which may in turn interfere with bone healing. Therefore, prophylaxis of fracture-associated pain is indispensable to postoperative comfort and satisfaction.

There is no denying the fact that pathologic pain is related to central glutaminergic system and N-methyl-d-aspartate (NMDA) receptor activation induced central sensitization. Also, we previously reported that neuroinflammation is associated with pain development and cognitive dysfunction. Ketamine, a NMDA receptor antagonist, is effective in reversing NMDA receptor activation underlying pain states. But the side effects of ketamine limit its clinical application, such as Delirium, gibberish and agitation. It is clarified that S-ketamine has lower side effects than ketamine and that antinociception of S-ketamine is stronger than ketamine. The following study is carried out to evaluate whether S-ketamine can prevent postoperative pain and cognitive impairment after tibial fracture and orthopedic surgery in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo tibial fracture with orthopedic surgery under a short general anesthesia of less than 2 hours
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.

Exclusion Criteria:

1. Subject has a diagnosis of bronchial asthma, coronary heart disease, severe hypertension, renal failure or liver failure.
2. Subject has a diagnosis of Insulin dependent diabetes.
3. Subject is allergy and contraindication to S-ketamine.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre- existing therapy with opioids.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.
7. Subject is obese (body mass index >30kg/m^2).
8. Subject is incapacity to comprehend pain assessment and cognitive assessment.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Mechanical hyperalgesia threshold on the palms of feet | 48 hours after surgery
  The mechanical hyperalgesia threshold was defined as the lowest force (g) necessary to bend a Von Frey filament, which was perceived to be painful by the patient and measured by Von Frey filament.

SECONDARY OUTCOMES:
Pain Score (NRS) | 48 hours after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Mechanical Hyperalgesia Threshold on the Dominant Inner Forearm | 48 hours after surgery
  The mechanical hyperalgesia threshold was defined as the lowest force (g) necessary to bend a Von Frey filament, which was perceived to be painful by the patient and measured by Von Frey filament
Time of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Total Dose of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Cumulative Sufentanyl Consumption | 48 hours after surgery
  Each patient was administered analgesics using a PCA (Patient-controlled analgesia) pump containing sufentanil (100μg) in normal saline at a total volume of 100 ml after leaving PACU (Postanesthesia care unit). This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5 ml with a 15-min lockout period. Sufentanyl cumulative consumption is recorded 48 hours postoperatively
Occurrence of Side Effects | 48 hours after surgery
  Occurrence of side effects: nausea, vomiting, dizziness, headache, shivering, pruritus
Mini-Mental State Examination (MMSE) | 48 hours after surgery
  Cognitive performance was assessed with Mini-Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Terrando N, Xu ZZ, Bang S, Jordt SE, Maixner W, Serhan CN, Ji RR. Distinct Analgesic Actions of DHA and DHA-Derived Specialized Pro-Resolving Mediators on Post-operative Pain After Bone Fracture in Mice. Front Pharmacol. 2018 May 1;9:412. doi: 10.3389/fphar.2018.00412. eCollection 2018. PMID 29765320
- [Background] Cui W, Li Y, Wang Z, Song C, Yu Y, Wang G, Li J, Wang C, Zhang L. Spinal caspase-6 regulates AMPA receptor trafficking and dendritic spine plasticity through netrin-1 in postoperative pain after orthopedic surgery for tibial fracture in mice. Pain. 2021 Jan;162(1):124-134. doi: 10.1097/j.pain.0000000000002021. PMID 32701657